CLINICAL TRIAL: NCT06357559
Title: Optical Coherence Tomography Angiography Changes in Choroidal Neovascularization in High Myopia
Brief Title: OCTA Changes in Choroidal Neovascularization in High Myopia
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Hamdy Abdelrahman, Dr., Sohag University
Other Study IDs: OCTA in Myopic CNV
Record Dates: First submitted 2024-03-11; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Myopic Choroidal Neovascularisation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OCTA — Optical Coherence Tomography Angiography

SUMMARY:
To Analyze the Ability of Optical Coherence Tomography Angiography ( OCT-A ) to detect the presence of myopic Choroidal Neovascularization and to describe the structural features of Myopic CNV..

DETAILED DESCRIPTION:
To Analyze the Ability of Optical Coherence Tomography Angiography ( OCT-A ) to detect the presence of myopic Choroidal Neovascularization and to describe the structural features of Myopic CNV.. regarding the size , shape , core , margin , Appearance , and activity of CNV..

ELIGIBILITY:
Inclusion Criteria:

* All Patients with High Myopia ( > -6 D or Axial Length > 26.5 mm ) with Fundoscopic Changes Consistent with CNVM , with Clear Media are Subjected to OCTA

Exclusion Criteria:

* Patients with Treated CNVs , or with other Causes of CNVs including :

Neovascular AMD , Idiopathic CNV , Traumatic , Inflammatory , Neoplastic , Degenerative ..

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with High Myopia ( Refractive Error > -6D or Axial Length > 26,5 mm ) with Fundoscopic Changes Consistent with CNVM.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Describing the Choroidal Neovascularization in High Myopic Patients diagnosed by OCTA | 1 year
  Describing the Choroidal Neovascularization in High Myopic Patients diagnosed by OCTA Regarding its Activity ..

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohno-Matsui K, Ikuno Y, Lai TYY, Gemmy Cheung CM. Diagnosis and treatment guideline for myopic choroidal neovascularization due to pathologic myopia. Prog Retin Eye Res. 2018 Mar;63:92-106. doi: 10.1016/j.preteyeres.2017.10.005. Epub 2017 Oct 28. PMID 29111299